CLINICAL TRIAL: NCT05188794
Title: Comparison of Two Different Approach Ultrasound Guided TAP Block on Pain Management of Laparoscopic Nephrectomy: Posterior or Lateral Approach?
Brief Title: Comparison of Two Different Approach TAP Block on Pain Management of Laparoscopic Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Serap Diker, Anaestesia and Reanimation Specialist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: E1-21-1814
Record Dates: First submitted 2021-11-22; First posted 2022-01-12 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Analgesia, Patient-Controlled; Postoperative Pain, Acute
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group L (Active Comparator): Lateral transversus abdominis plane(TAP) block
  Interventions: Procedure: lateral tap block
- Group P (Active Comparator): Posterior transversus abdominis plane block
  Interventions: Procedure: posterior tap block

INTERVENTIONS:
Procedure: lateral tap block — In the axial plane on the midaxillary line between the subcostal margin and the iliac crest with a linear probe using a 12 cm insulated nerve block needle is advanced in planely from skin, external, and internal oblique muscles to the target of fascial plane between the internal oblique and the transversus abdominis muscles.
  Arms: group L
Procedure: posterior tap block — In the axial plane on the midaxillary line a linear probe using a 12 cm insulated nerve block needle is advanced posteriorly to the most posterior limit of the TAP between the internal oblique and transversus abdominis muscles.
  Arms: Group P

SUMMARY:
Primary aim is to compare the effectiveness of the posterior approach Transversus abdominis plane block (P-TAP) and the lateral approach Transversus abdominis plane block (L-TAP) technique on the pain management of the laparoscopic nephrectomy in terms of visual analog pain scale and postoperative opioid consumption. Secondary aim is to compare complication rates of the two techniques.

DETAILED DESCRIPTION:
Patients included in the study will be randomized into two groups (group L and group P) in the preoperative period. Following routine anesthesia induction TAP block will be applied to group L patients with the lateral approach technique, and to group P patients with the posterior approach technique. Regional block complications will be recorded.

Standard laparoscopic nephrectomy surgical method will be applied. 1g of paracetamol and 4mg of dansetron will be administered to both groups 15 minutes before the end of the operation. The pain intensity of the patients will be questioned and VAS values will be recorded at 0, 1, 2, 6, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASAI-III patients undergoing laparoscopic nephrectomy
* 18<BMI<40

Exclusion Criteria:

* infection at the block site
* coagulation disorder
* pregnancy
* kidney failure
* liver failure
* heart failure
* allergy to local anesthetics
* patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Visual analog pain scale 0 | at the PACU arrival
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual analog pain scale 1 | Postoperative first hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual Analog Pain scale 2 | Postoperative second hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual analog pain scale 6 | Postoperative sixth hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual Analog Pain scale 12 | Postoperative 12. hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual Analog Pain scale 18 | Postoperative18. hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
Visual Analog Pain scale 24 | Postoperative 24. hour
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.
opioid comsuption | Within 24 hours postoperatively
  Patients will be asked about the severity of pain. They will be told that 0 = no pain, 10 = severe pain, and they will be asked to determine a number between 0 and 10 for the severity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: MİYASE SERAP DİKER, DOCTOR, Principal Investigator — ANKARA CİTY HOSPİTAL
Locations (1):
- Ankara City Hospital,Bilkent, Ankara, Cankay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No